CLINICAL TRIAL: NCT03309592
Title: Investigator Sponsored Research Proposal : Efficacy and Safety of Combination Ambrisentan and TadaLafil in PATiEnts With PortoPulmonary Hypertension (ESCALATE-PPH)
Brief Title: Efficacy and Safety of Combination Ambrisentan and Tadalafil in Patients With Portopulmonary Hypertension
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of eligible participants and failure to meeting study enrollment.
Sponsor: Ochsner Health System (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESCALATE-PPH
Record Dates: First submitted 2017-06-05; First posted 2017-10-13 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Portopulmonary Hypertension; Pulmonary Hypertension; Cirrhosis, Liver
MeSH Terms: conditions — Hypertension, Pulmonary; Liver Cirrhosis | interventions — ambrisentan; Tadalafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combination Therapy (Other): Qualifying participants will begin combination therapy with ambrisentan pill 5 mg daily and tadalafil pill 20 mg. After one week of therapy, patients will increase tadalafil pill to 40 mg daily and continue ambrisentan pill 5 mg daily. On day 15, patients will increase ambrisentan pill to 10 mg daily and continue at 40 mg of tadalafil pill daily.
  Interventions: Drug: Ambrisentan Pill; Drug: Tadalafil Pill

INTERVENTIONS:
Drug: Ambrisentan Pill — Will be administered as stated in Arm/Group Descriptions
  Other Names: Letairis
Drug: Tadalafil Pill — Will be administered as stated in Arm/Group Descriptions
  Other Names: Adcirca

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of the combination of ambrisentan and tadalafil in reducing mPAP to below 35mmHg in patients with moderate to severe Portopulmonary Hypertension (POPH) as a means to candidacy for liver transplantation.

DETAILED DESCRIPTION:
The outcome of liver transplantation (LT) in the presence of moderate to severe POPH is significantly poor with a 50% reported mortality rate in LT recipients having a mean pulmonary artery pressure (mPAP) >35 mmHg and 100% when the mPAP is greater than 50 mmHg; therefore, making moderate to severe POPH a contraindication to liver transplants. Those recipients with significant pulmonary artery pressure (PAP) may be denied the opportunity for transplant unless the mPAP is brought below 35 mmHg with medical treatment. This study will test the efficacy & safety of the combination of using ambrisentan and tadalfil in reducing the Pulmonary Arterial Pressure to below 35 mmHg in patients with moderate to severe POPH as a means to candidacy for liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Child-Pugh Class Class A & B Cirrhosis
* mPAP ≥35mmHg
* Pulmonary Capillary Wedge Pressure (PWCP) <15mmHg on Right Heart Catheterization's (RHCs)
* mPAP > 50mmHg will be considered eligible unless they are World Health Organization (WHO) Functional Class IV

Exclusion Criteria:

* End stage renal disease on hemodialysis (ESRD on HD)
* Renal dysfunction and GFR < 30
* AST, ALT > 5 times the upper limit of normal
* Total bilirubin ≥ 6.0
* INR > 2

  * Initially, Child-Pugh Class C patients will be excluded; however, after the first 5 patients are included, if there is no signal of worsening liver function, the protocol may be amended to include patients with Class C cirrhosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Reduction in mPAP to 35mmHg | 2 months post initiation of therapy
  A Right Heart Catheterization will be performed in order to see if there's a reduction in mPAP to less than 35mmHg from baseline

SECONDARY OUTCOMES:
Blood Pressure | 2 months post therapy
  Systemic Blood pressure
mPAP Reduction | 2 months post initiation of therapy
  Percent reduction in mPAP will be assessed and measured from baseline via RHC
Post-Transplant Survival Outcome: Alive or Dead at 30 days | Post-op Day 1 and 30
  Post-transplant survival comparing subjects with or without history of POPH
Kidney function evaluation through measurement of Creatinine levels (mg/dL) | baseline, 1 month, 2 month, 3 month, 6 month, 9 month, 12 months/end of treatment, 1 month post transplant
  Comprehensive metabolic panel will be completed at 2 months post therapy to assess kidney function
Liver Function test measured by AST (iu/L) | baseline, 1 month, 2 month, 3 month, 6 month, 9 month, 12 months/end of treatment, 1 month post transplant
  AST will be done to monitor and measure the degree of cirrhosis on the liver as well as the overall function of the liver
Liver Function test measured by ALT (iu/L) | baseline, 1 month, 2 month, 3 month, 6 month, 9 month, 12 months/end of treatment, 1 month post transplant
  ALT test will be done to monitor and measure the degree of cirrhosis on the liver as well as the overall function of the liver
Liver Function test measured by Bilirubin (mg/dL) | baseline, 1 month, 2 month, 3 month, 6 month, 9 month, 12 months/end of treatment, 1 month post transplant
  Bilirubin test will be done to monitor and measure the degree of cirrhosis on the liver as well as the overall function of the liver
Liver Function test measured by INR | baseline, 1 month, 2 month, 3 month, 6 month, 9 month, 12 months/end of treatment, 1 month post transplant
  INR test will be done to monitor and measure the degree of cirrhosis on the liver as well as the overall function of the liver
Right Ventricular (RV) Size in centimeters | Baseline, 1-month, 6-month and 12 months post therapy, 1 month post transplant
  To measure Right Ventricular Size in centimeters
Right Ventricular (RV) Qualitative Systolic Function: assessment that is categorized as normal, mildly depressed, moderately depressed or severely depressed | Baseline, 1-month, 6-month and 12 months post therapy, 1 month post transplant
  To measure Right Ventricular Qualitative Systolic Function assessment that is categorized as normal, mildly depressed, moderately depressed or severely depressed
Right Ventricular (RV) Function in centimeters | Baseline, 1-month, 6-month and 12 months post therapy and 1-month post transplant
  Tricuspid Annular Plane Systolic Excursion (TAPSE) measured in centimeters
Biomarker of Right ventricular failure | baseline, 1 month, 2 month, 3 month, 6 month, 9 month, 12 months/end of treatment, 1 month post transplant
  serum BNP
New York Heart Association Functional class | baseline, 1 month, 2 month, 3 month, 6 month, 9 month, 12 months/end of treatment, 1 month post transplant
  NYHA FC will be assessed by clinician at baseline and each subsequent visit
Change in 6 Minute Walk Distance | baseline, 1 month, 2 month, 3 month, 6 month, 9 month, 12 months/end of treatment, 1 month post transplant
  6 Minute walk will be performed at baseline and each study visit

CONTACTS AND LOCATIONS:
Overall Officials: Stacy Mandras, MD, Principal Investigator — Director, Pulmonary Hypertension
Locations (1):
- Ochsner Clinic Foundation, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No